CLINICAL TRIAL: NCT03247764
Title: A Registration Study on Drug Treatment for Comorbid Depression in Patients With Epilepsy in East China
Brief Title: A Registration Study on Depression in Patients With Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Regist-EP and DP
Record Dates: First submitted 2017-08-03; First posted 2017-08-14 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Epilepsy; Depression
Keywords: epilepsy; depression; drug treatment
MeSH Terms: conditions — Epilepsy; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with the comorbidity of epilepsy and depression: the clinical data, psychological assessment, and drug treatments will be investigated in patients with the comorbidity of epilepsy and depression

INTERVENTIONS:
Other:  — observational study

SUMMARY:
The aim of this study is to register the drug treatment of depression in patients with epilepsy in East China.

DETAILED DESCRIPTION:
As the treatment rate for depression in epilepsy is unclear and the discordant voice of choosing antidepressants for most doctors, this prospective observational cohort study was designed to better understand the current situation of drug treatments in patients with the comorbidity of epilepsy and depression in East China. The secondary outcome was to investigate whether baseline depressive symptoms had an influence on seizure-control in patients with epilepsy at follow-up.

ELIGIBILITY:
The inclusion criteria were as follows: (1) age 18-75, no gender limited; (2) diagnosis of epilepsy according to the definition by ILAE in 2014; (3) the score of 17-item Hamilton Depression Rating Scale greater than 7; (4) Obtaining informed consent of participants. The exclusion criteria were any of the following: (1) having psychiatric symptoms such as hallucination or delusion; (2) progressive neurological diseases and malignant tumors; (3) severe cognitive dysfunction (the score of MMSE less than 10).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with the comorbidity of epilepsy and depression present to the neurology department at 8 tertiary hospitals in East China
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
the drug treatment rate of depression in patients with epilepsy | 6 months
  the drug treatment rate at baseline and 6 months at follow-up

SECONDARY OUTCOMES:
the influence of depression on seizure-control | 6 months
  whether depression at baseline affects seizure-control 6 months later

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, PhD, Principal Investigator — Fudan University
Locations (7):
- China (7):
  - Department of Neurology, Huashan Hospital, Fudan University, Shanghai, China, Shanghai, Shanghai Municipality
  - Department of Neurology, Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Anhui Provincial Hospital, Hefei
  - Nanjing Brain Hospital, Nanjing
  - Shanghai General Hospital, Shanghai
  - The Second Affiliated Hospital of Suzhou University, Suzhou
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou